CLINICAL TRIAL: NCT05310669
Title: Inspiratory Effort Assessed Through Nasal Pressure Measurement in Patients With Idiopathic Pulmonary Fibrosis
Acronym: NASA
Status: Recruiting | Type: Observational
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Roberto Tonelli, Principal investigator, University of Modena and Reggio Emilia
Other Study IDs: UModenaReggio16
Record Dates: First submitted 2022-03-25; First posted 2022-04-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Fibrosis, Pulmonary
Keywords: Inspiratory effort; Lung Damage; Fibrosis progression
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Nasal pressure assessment — Once the patient is enrolled nasal pressure will be measured through a dedicated pressure line located at the nostril entrance and connected to a dedicated pressure transducer (OptiVentTM, SIDAM, Mirandola, Italy). Measured nasal pressure will be the result of the variation between inspiratory and expiratory pressure (DeltaPnose).

SUMMARY:
Idiopathic Pulmonary Fibrosis (IPF) is a fibrosing progressive interstitial lung disease with unknown etiology, with a median survival of 3 years since first diagnosis. The typical radiologic pattern of the disease is usual interstitial pneumonia (UIP) defined by basal and peripheral (subpleural) predominance and a typical cystic degeneration of lung parenchyma (honeycombing), interstitial fibrotic thickening and traction bronchiectasis. Despite the recent introduction of two antifibrotic treatments (Pirfenidone and Nintendanib) which proved to be successful in slowing the decline of pulmonary function in patients with IPF, a benefit of these therapies on average survival remains yet to be demonstrated.

A significant part of patients affected by IPF die due to progressive worsening of respiratory failure, often accelerated by the insurgence of acute events, like acute exacerbations. Processes leading to the development and progression of IPF are not yet completely understood. We might hypothesize a regenerative deficit in the lungs of subjects affected, due to a dysregulation of repair mechanism in response to repeated damage (inflammatory, mechanics, infectious, chemical) to the alveolar and vascular epithelium. Moreover, mechanism of damage caused by aging in tissues, with a dysfunction in resident stem cell, might contribute to progression. Patients with IPF undergo mechanical alterations of respiratory system due to progressive restrictive deficit caused by reduction in total lung capacity. This functional alteration generates an ineffective and superficial ventilation due to the waste of the majority inspiratory effort spent in ventilating dead anatomical space. When physical effort occurs, the increased ventilatory necessity and the inability to compensate due to functional impairment leads to increased inspiratory effort and subsequent increase in negative intrathoracic pressure. Recent studies have demonstrated how exerting a pressure (for example when the patient is mechanically ventilated) on lung tissue of subjects with IPF and UIP pattern can generate damage due to unfavorable mechanism of mechanotransduction caused by the pathological behavior of fibrotic lung (''squishy ball lung''). Studies investigating inspiratory effort during spontaneous breathing and respiratory failure highlighted how negative values of intrathoracic pressure might induce self induced lung injury.

Respiratory effort can be quantified measuring esophageal pressure through a pressure transducer inserted with a nasogastric tube in the inferior third part of the esophagus. Measuring esophageal pressure is a precise and accurate way of quantifying inspiratory effort, however its use in daily clinical practice is limited by invasiveness of the maneuver, high cost and need for specific clinical training. Physiological studies show that nasal pressure measured at the entrance of the nostril might correlate with esophageal pressure and therefore estimate inspiratory effort of the patient in a noninvasive way.

The goal of our study is to evaluate the role of respiratory effort during spontaneous breathing as a potential source of mechanical damage (hence favoring disease progression) in subjects with IPF and UIP pattern. The study aims to identify patient with an unfavorable mechanical phenotype defined by the simultaneous presence of UIP pattern and elevated inspiratory effort after physical activity.

ELIGIBILITY:
Inclusion Criteria:

Patients treated in Center for Rare diseases of Azienda Ospedaliero-Universitaria Policlinico di Modena will be considered eligible if satisfying the following inclusion criteria:

* Patient with IPF and UIP pattern
* Need for radiological evaluation through HRCT

Exclusione criteria

* Age below 18
* Pregnancy
* Inability to sign informed consent
* COPD
* Neuromuscular diseases
* Evidence of IPF acute exacerbation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Center for Rare diseases of Azienda Ospedaliero-Universitaria Policlinico di Modena, Italy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Inspiratory effort | 2 hours.
  Quantification of inspiratory effort through nasal pressure before and after physical activity will be therefore considered as primary exploratory outcome.

SECONDARY OUTCOMES:
Forced expiratory volume decline | 6 months
  Change in forced expiratory volume at 6 months will be correlated with values of respiratory effort

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Policlinico di Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: Undecided